CLINICAL TRIAL: NCT03923582
Title: Training for Health Professionals in Tanzania
Acronym: THP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other); Johns Hopkins University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00006904; R01HD092655 (NIH)
Record Dates: First submitted 2018-08-01; First posted 2019-04-22 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Health Knowledge, Attitudes, Practice; Training
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: Development and testing of a sexual health curriculum for Midwifery, Nursing and Medical Students.
Who Masked: Outcomes Assessor
Masking Description: A randomized, controlled, single blinded trial, stratified by health profession, of the intervention vs waitlist control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): A four-day comprehensive sexual health curriculum tailored for Africa.
  Interventions: Behavioral: Comprehensive sexual health curriculum
- Waitlist control (No Intervention): Participants in this arm completed a follow-up survey and were scheduled to receive the intervention after the end of the trial.

INTERVENTIONS:
Behavioral: Comprehensive sexual health curriculum — This is a randomized, controlled, single blinded, trial, stratified by health profession, of the intervention versus waitlist control assessing knowledge, attitude change and skill development. At the end of the intervention as compared with waitlist controls.
  The intervention was a 4-day, Afrocentric, comprehensive sexual health curriculum. Tanzanian faculty wrote the curriculum in English and Kiswahili to address the most common sexual health challenges clinicians experience in Tanzania. The 4-day curriculum covers sexual health across the lifespan, LGBT and sexual violence, clinical skills training, ethics and policy writing, and community resources and cultural considerations.
  Arms: Intervention Arm

SUMMARY:
The goal of this randomized, controlled, single blinded trial is to evaluate the effectiveness of an Afrocentric sexual health curriculum on health professional students' knowledge, attitudes, and clinical skills in providing sexual health care in Tanzania.

DETAILED DESCRIPTION:
There were 563 students recruited for the study that met the eligibility requirement. A total of 412 students gave consent and were randomized into intervention and control groups. At baseline, participants took a survey covering demographic information, educational background, sexual health knowledge, and attitudes toward sexual health topics. After completing the survey, participants participated in two standardized patient interviews involving actors role playing sexual health-related patient scenarios.

Those who were in the intervention arm participated in a 4-day sexual health curriculum followed by a post-test survey measuring sexual health knowledge, attitudes, and evaluation of sexual health training.

Three to four months later, intervention and waitlist control participants completed a follow-up survey assessing sexual health knowledge and attitudes toward sexual health topics and standardized patients scenarios.

Multiple linear regression was used to assess the overall effectiveness of the sexual health curriculum on the attitudes, knowledge, and skills of health professionals after it has been implemented.

ELIGIBILITY:
Inclusion Criteria:

1. current student at MUHAS in midwifery, nursing, or medicine.
2. 3rd or 4th year for medical students or 2nd or 3rd year for nursing and midwifery students.
3. able to attend the full 4-day training during the first week of student vacation.
4. fluent in English (the language of instruction at MUHAS) and Kiswahili (the lingua franca in Tanzania).
5. willing to volunteer and complete all evaluation procedures.

Exclusion Criteria:

1. students who will not be able to attend MUHAS all days of the seminar or be on the MUHAS campus for the follow-up dates.
2. students who express severe reservations about attending (e.g., due to religious objections).
3. Students who express fear of violence due to attending (e.g., from a spouse or relative).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2022-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: B.R Simon Rosser, PhD, Principal Investigator — University of Minnesota
Locations (2):
- University of Minnesota, Minneapolis, Minnesota, United States
- Muhimbili University of Health and Allied Sciences (MUHAS), Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: No
Only group data will be analyzed.

REFERENCES:
- [Background] Ross MW, Leshabari S, Rosser BRS, Trent M, Mgopa L, Wadley J, Kohli N, Agardh A. Evaluation of an assessment instrument for a sexual health curriculum for nurses and midwifery students in Tanzania: The sexual health education for professionals scale (SHEPS). Appl Nurs Res. 2018 Apr;40:152-156. doi: 10.1016/j.apnr.2018.01.005. Epub 2018 Feb 1. PMID 29579491
- [Background] Rosser BRS, Mgopa L, Leshabari S, Ross MW, Lukumay GG, Massawe A, Mkonyi E, Mohammed I, Mushy S, Mwakawanga D, Trent M, Wadley J. Legal and Ethical Considerations in the Delivery of Sexual Health Care in Tanzania. Afr J Health Nurs Midwifery. 2020;3(7):84-102. Epub 2020 Dec 27. PMID 34723251
- [Background] Mgopa LR, Rosser BRS, Ross MW, Lukumay GG, Mohammed I, Massae AF, Leshabari S, Mkonyi E, Mushy SE, Mwakawanga DL, Trent M, Wadley J, Bonilla ZE. Cultural and clinical challenges in sexual health care provision to men who have sex with men in Tanzania: a qualitative study of health professionals' experiences and health students' perspectives. BMC Public Health. 2021 Apr 7;21(1):676. doi: 10.1186/s12889-021-10696-x. PMID 33827508
- [Background] Mgopa LR, Ross MW, Lukumay GG, Mushy SE, Mkony E, Massae AF, Mwakawanga DL, Leshabari S, Mohamed I, Trent M, Wadley J, Bonilla ZE, Rosser BRS. Perceptions of Sexual Healthcare Provision in Tanzania: a Key Informant Qualitative Study. Sex Res Social Policy. 2022 Sep;19(3):849-859. doi: 10.1007/s13178-021-00607-5. Epub 2021 Jul 3. PMID 36172532
- [Background] Mgopa LR, Rosser BRS, Ross MW, Mohammed I, Lukumay GG, Massae AF, Mushy SE, Mwakawanga DL, Mkonyi E, Trent M, Bonilla ZE, Wadley J, Leshabari S. Clinical Care of Victims of Interpersonal Violence and Rape in Tanzania: A Qualitative Investigation. Int J Womens Health. 2021 Jul 24;13:727-741. doi: 10.2147/IJWH.S301804. eCollection 2021. PMID 34335058
- [Background] Mushy SE, Rosser BRS, Ross MW, Lukumay GG, Mgopa LR, Bonilla Z, Massae AF, Mkonyi E, Mwakawanga DL, Mohammed I, Trent M, Wadley J, Leshabari S. The Management of Masturbation as a Sexual Health Issue in Dar es Salaam, Tanzania: A Qualitative Study of Health Professionals' and Medical Students' Perspectives. J Sex Med. 2021 Oct;18(10):1690-1697. doi: 10.1016/j.jsxm.2021.07.007. Epub 2021 Aug 24. PMID 34452866
- [Background] Mwakawanga DL, Mkonyi E, Mushy SE, Trent M, Bonilla Z, Massae AF, Lukumay GG, Mgopa LR, Mohammed I, Wadley J, Ross MW, Leshabari S, Rosser BRS. Would you offer contraception to a 14-year-old girl? Perspectives of health students and professionals in Dar es Salaam, Tanzania. Reprod Health. 2021 Dec 11;18(1):245. doi: 10.1186/s12978-021-01294-6. PMID 34895267
- [Background] Mkonyi E, Mwakawanga DL, Rosser BRS, Bonilla ZE, Lukumay GG, Mohammed I, Mushy SE, Mgopa LR, Ross MW, Massae AF, Trent M, Wadley J. The management of childhood sexual abuse by midwifery, nursing and medical providers in Tanzania. Child Abuse Negl. 2021 Nov;121:105268. doi: 10.1016/j.chiabu.2021.105268. Epub 2021 Aug 17. PMID 34416472
- [Background] Lukumay GG, Mgopa LR, Mushy SE, Rosser BRS, Massae AF, Mkonyi E, Mohammed I, Mwakawanga DL, Trent M, Wadley J, Ross MW, Bonilla Z, Leshabari S. Community myths and misconceptions about sexual health in Tanzania: Stakeholders' views from a qualitative study in Dar es Salaam Tanzania. PLoS One. 2023 Feb 10;18(2):e0264706. doi: 10.1371/journal.pone.0264706. eCollection 2023. PMID 36763616
- [Background] Rosser BRS, Mkoka DA, Rohloff CT, Mgopa LR, Ross MW, Lukumay GG, Mohammed I, Massae AF, Mkonyi E, Mushy SE, Mwakawanga DL, Kohli N, Trent ME, Wadley J, Bonilla ZE. Tailoring a sexual health curriculum to the sexual health challenges seen by midwifery, nursing and medical providers and students in Tanzania. Afr J Prim Health Care Fam Med. 2022 May 31;14(1):e1-e9. doi: 10.4102/phcfm.v14i1.3434. PMID 35695444
- [Derived] Rosser BRS, Kohli N, Bates AJ, Talley KMC, Wright MM, Polter EJ, Wheldon CW, Haggart R, Dickstein DR, Ross MW, Zhang Z, West W, Konety BR. Does sexual rehabilitation work for gay and bisexual prostate cancer patients? Acceptability, feasibility, and efficacy results from the Restore-2 randomized controlled trial. J Cancer Surviv. 2024 Sep 12. doi: 10.1007/s11764-024-01672-6. Online ahead of print. PMID 39266938
- [Derived] Mushy SE, Mkoka DA, Lukumay GG, Massae AF, Rohloff CT, Mgopa LR, Mwakawanga DL, Kohli N, Ross MW, Mkonyi E, Trent M, Athumani K, Kulasingam S, Rosser BRS. The need for and acceptability of a cancer training course for medical and nursing students in Tanzania: a convergent mixed methods study. BMC Med Educ. 2024 Jun 3;24(1):614. doi: 10.1186/s12909-024-05497-w. PMID 38831409

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Arm: A four-day comprehensive sexual health curriculum tailored for Africa.
  Comprehensive sexual health curriculum: This is a randomized, controlled, single blinded, trial, stratified by health profession, of the intervention versus waitlist control assessing knowledge, attitude change and skill development. At the end of the intervention as compared with waitlist controls.
  The intervention was a 4-day, Afrocentric, comprehensive sexual health curriculum. Tanzanian faculty wrote the curriculum in English and Kiswahili to address the most common sexual health challenges clinicians experience in Tanzania. The 4-day curriculum covers sexual health across the lifespan, LGBT and sexual violence, clinical skills training, ethics and policy writing, and community resources and cultural considerations.
Period: Overall Study
Arm/Group | Intervention Arm | Waitlist Control
Started | 206 | 206
Completed | 203 | 205
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Waitlist Control | Total
Number analyzed (Participants) | 206 | 206 | 412
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.90 (2.36) | 24.05 (2.56) | 24 (2.46)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 64 | 62 | 126
  Male | 137 | 139 | 276
  Other/Prefer not to answer | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 206 | 206 | 412
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Sexual Health Knowledge [Mean (Standard Deviation); unit: units on a scale] | 6.170 (2.113) | 6.427 (2.091) | 6.299 (2.103)
Sexual Health Knowledge: Confidence in Ability to Discuss [Mean (Standard Deviation); unit: units on a scale] | 153.485 (20.632) | 152.8452 (21.349) | 153.165 (20.970)
Sexual Health Attitudes: Confidence in Having Knowledge [Mean (Standard Deviation); unit: units on a scale] | 150.141 (24.430) | 150.704 (24.511) | 150.422 (24.442)
Sexual Counseling Skills: Interpersonal Communications [Mean (Standard Deviation); unit: units on a scale] | 22.583 (4.198) | 21.951 (4.403) | 22.267 (4.308)
Sexual Counseling Skills: Medical History Taking [Mean (Standard Deviation); unit: units on a scale] | 6.019 (2.419) | 6.029 (2.397) | 6.024 (2.405)
Sexual Health Belief [Mean (Standard Deviation); unit: units on a scale] | 79.825 (9.292) | 78.320 (9.555) | 79.073 (9.443)

OUTCOME MEASURES:

1. Primary Outcome: Change in Sexual Health Knowledge Score From Baseline to Follow-up
Description: Sexual health knowledge was assessed using 16 multichoice items created by the research team. The items covered female sexual health concerns (2 items), sexual development and masturbation (3 items), sexual orientation (3 items), sexual violence (3 items), sexuality in middle age (3 items), sexual history taking and sexual counseling (2 items). Total scores were used for analysis (maximum total score of 16). Participants get one point for every item they answer correctly. Because there are 16 items in this section, participants can have a minimum total score of 0 and a maximum total score of 16. A higher score signifies better sexual health knowledge. A single value was calculated for the intervention arm and waitlist control from difference scores (calculated as follow-up minus baseline scores).
Time Frame: At Baseline and 3-4 months Follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Waitlist Control
Number analyzed (Participants) | 198 | 198
score on a scale | 3.551 (2.310) | 0.086 (2.341)

2. Primary Outcome: Change in Sexual Health Attitudes: Confidence in Ability to Discuss From Baseline to Follow-up
Description: Confidence in their ability to discuss the sexual health of patients, and confidence in their ability to discuss their patients' sexual health concerns were assessed using the Sexual Health Education for Professionals Scale (SHEPS). This section consists of 37 items where participants rate their confidence from (1) very unconfident to (5) confident. Because there are 37 items in this section, participants can have a minimum total score of 37 and a maximum total score of 185. A higher value signifies better confidence in the ability to discuss sexual health topics. A single value was calculated for the intervention arm and waitlist control from difference scores (calculated as follow-up minus baseline scores).
Time Frame: At Baseline and 3-4 months Follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Waitlist Control
Number analyzed (Participants) | 198 | 198
score on a scale | 19.389 (20.517) | -2.449 (19.036)

3. Primary Outcome: Change in Sexual Health Attitudes: Confidence in Having Knowledge From Baseline to Follow-up
Description: Confidence in their knowledge to assess the sexual health of patients, and confidence in their ability to discuss their patient's sexual health concerns were assessed using the Sexual Health Education for Professionals Scale (SHEPS). This section consists of 37 items where participants rate their confidence from (1) very unconfident to (5) confident. Because there are 37 items in this section, participants can have a minimum total score of 37 and a maximum total score of 185. A higher value signifies better confidence in having knowledge of sexual health topics. A single value was calculated for the intervention arm and waitlist control from difference scores (calculated as follow-up minus baseline scores).
Time Frame: At Baseline and 3-4 months Follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Waitlist Control
Number analyzed (Participants) | 198 | 198
score on a scale | 22.768 (23.983) | -4.242 (20.780)

4. Primary Outcome: Change in Sexual Counseling Skills: Interpersonal Communications From Baseline to Follow-up
Description: Skills were assessed by faculty raters assessing two videos (per each time point) of student counseling blind to whether the participant was in the intervention or control group and whether the assessment was at baseline or follow-up. Each participant was rated on 10 items assessing their interpersonal communication (IC) abilities. Each item was on a 3-point scale (0=not done; 1=partially done; 2=done). The scale has a minimum score of 0 and a maximum score of 20 per video. We aggregated scores for each time point by summing the two videos at each time point. Therefore, the minimum total score is 0 and the maximum total score is 40. A higher score value signifies better interpersonal communication skills. A single value was calculated for the intervention arm and waitlist control from difference scores based on the sum of the scores at baseline and the sum of the scores at followup.
Time Frame: At Baseline and 3-4 months Follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Waitlist Control
Number analyzed (Participants) | 198 | 198
score on a scale | 6.890 (6.247) | -0.975 (5.831)

5. Primary Outcome: Change in Sexual Counseling Skills: Medical History Taking From Baseline to Follow-up
Description: Skills were assessed by faculty raters assessing the two videos (per time point) of student counseling blind to whether the participant was in the intervention or control group and whether the assessment was at baseline or follow-up. Medical history taking (MHT) was rated by six key pieces of information on a 2-point scale, where 0=not obtained information and 1=obtained information. The scale has a minimum score of 0 and a maximum score or 6 per video. We aggregated scores for each time point by summing the two videos at each time point. Therefore, the minimum total score is 0 and the maximum total score is 12. A higher score value signifies better medical history taking skills. A single value was calculated for the intervention arm and waitlist control from difference scores based on the sum of the scores at baseline and the sum of the scores at followup.
Time Frame: At Baseline and 3-4 months Follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Waitlist Control
Number analyzed (Participants) | 198 | 198
score on a scale | 1.828 (2.905) | -0.682 (2.688)

6. Primary Outcome: Change in Sexual Health Beliefs From Baseline to Follow-up
Description: The SHEPS Attitudes section comprises 27 items. Participants rate their level of agreement (1=strongly agree; 5=strongly disagree), with 13 items being reverse coded. Because there are 27 items in this section, participants can have a minimum total score of 27 and a maximum total score of 135. Low scores correspond to "liberal" views and high scores correspond to "conservative" views. A single value was calculated for the intervention arm and waitlist control from difference scores (calculated as follow-up minus baseline scores).
Time Frame: At Baseline and 3-4 months Follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Waitlist Control
Number analyzed (Participants) | 198 | 198
score on a scale | -11.106 (11.595) | -0.929 (8.755)

ADVERSE EVENTS:
Description: adverse events were not collected
Arm/Group | Intervention Arm | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT03923582/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT03923582/SAP_001.pdf